CLINICAL TRIAL: NCT05174013
Title: A Randomised, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics, Target Engagement and Immunogenicity of a Single Subcutaneous Dose of GSK3858279 Administered to Healthy Caucasian, Chinese and Japanese Participants
Brief Title: Safety, Tolerability, Pharmacokinetics and Target Engagement of GSK3858279 in Healthy Caucasian, Chinese and Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 212979
Record Dates: First submitted 2021-12-22; First posted 2021-12-30 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pain
Keywords: Pharmacokinetics; Safety; Tolerability; GSK3858279; Placebo; Caucasian; Chinese; Japanese
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This will be a double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- GSK3858279 Caucasian (Experimental): Participants received 240 milligrams (mg) of GSK3858279 administered as separate subcutaneous (SC) injection to healthy Caucasian participants.
  Interventions: Drug: GSK3858279
- GSK3858279 Chinese (Experimental): Participants received 240 mg of GSK3858279 administered as separate SC injection to healthy Chinese participants.
  Interventions: Drug: GSK3858279
- GSK3858279 Japanese (Experimental): Participants received 240 mg of GSK3858279 administered as separate SC injection to healthy Japanese participants.
  Interventions: Drug: GSK3858279
- Caucasian Placebo (Placebo Comparator): Participants received single dose of Placebo administered as separate SC injection to healthy Caucasian participants.
  Interventions: Drug: Placebo
- Chinese Placebo (Placebo Comparator): Participants received Single dose of Placebo administered as separate SC injection to healthy Chinese participants.
  Interventions: Drug: Placebo
- Japanese Placebo (Placebo Comparator): Participants received Single dose of Placebo administered as separate SC injection to healthy Japanese participants.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK3858279 — GSK3858279 will be administered
  Arms: GSK3858279 Caucasian; GSK3858279 Chinese; GSK3858279 Japanese
Drug: Placebo — Placebo will be administered
  Arms: Caucasian Placebo; Chinese Placebo; Japanese Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), target engagement (TE) and immunogenicity of GSK3858279 when administered to healthy Caucasian, Chinese and Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants between 20 and 65 years of age inclusive, at the time of signing the informed consent.
* Volunteers who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Participant capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Participants who have evidence of completed vaccination for Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) with an approved vaccine.
* Body weight within the range 45 - 100 killogram (kg) and body mass index (BMI) within the range 18-29.9 kg per meter square (/m2) (inclusive).
* Japanese participants are eligible based on meeting all of the following:
* Participants born in Japan
* Descendants of four ethnic Japanese grandparents and two ethnic Japanese parents.
* Have lived outside Japan for less than (<) 10 years at the time of screening
* Chinese participants are eligible based on meeting all of the following
* Participants born in mainland China, Hong Kong or Taiwan
* Descendants of four Chinese grandparents and two Chinese parents
* Have lived outside China, Hong Kong or Taiwan for <10 years at the time of screening
* Caucasian participants are eligible based on meeting the following
* Declaration of familial Caucasian/European ancestry (having 2 parents of Caucasian/European ancestry and 4 grandparents of Caucasian/European ancestry)
* Male or female participant
* Male participants are eligible to participate if they agree to the following for at least 28 weeks after the dose of study intervention: Refrain from donating sperm plus either be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent OR must agree to use contraception/barrier as detailed below: agree to use a male condom and should also be advised of the benefit for a female partner to use a highly effective method of contraception as a condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant.
* A female participant is eligible to participate if she is of non-reproductive potential.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* Personal or family history of cardiomyopathy.
* Abnormal blood pressure at screening as determined by the investigator.
* History of symptomatic herpes zoster.
* Evidence of active or latent tuberculosis (TB) as documented by medical history, examination, and TB testing with a positive (not indeterminate) QuantiFERON test.
* Significant allergies to humanized monoclonal antibodies as per principal investigator's and GSK medical monitor's judgements.
* History or evidence of clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* History of lymphoma, leukaemia, or any malignancy within the last 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years.

ALT greater than (>)1.5 times upper limit of normal (ULN) .

* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Corrected QT (QTc) >450 milliseconds (msec).
* History of Stevens Johnson Syndrome.
* Known immunodeficiency.
* Participants with a chronic infection (for example [e.g.], osteomyelitis), who have been receiving treatment within three months prior to dosing or individuals with an active infection.
* Previous or current history of bleeding diathesis, excessive bleeding or coagulation disorders.
* History of significant medical illness in the opinion of the investigator would interfere with the study procedures and / or assessments.
* Intended use of over-the-counter or prescription medication including herbal medications within 7 days prior to dosing until final follow-up visit.
* Live vaccine(s) or plans to receive such vaccines within 1 month of screening until final follow-up visit.
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing.
* Treatment with antiplatelet or anticoagulant agents within 7 days of dosing.
* Major surgery (as per investigator's judgement) within 3 months prior to dosing.
* Participation in the study would result in loss of blood or blood products in excess of 500 milliliters (mL) within 3 months.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrolment or past participation in any other clinical study involving an investigational drug intervention within the last 3 months or 5 half-lives (whichever is longer) of signing the ICF.
* Presence of Hepatitis B surface antigen (HBsAg) at screening.
* Presence of the Hepatitis B core antibody (HBcAb) at screening.
* Positive Hepatitis C antibody test result at screening.
* Positive Hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* Abnormal clinically significant echocardiogram at screening, as assessed by the investigator.
* Cardiac troponin or N-terminal pro B-type natriuretic peptide (NT-proBNP) levels out of normal range at screening.
* Positive pre-study drug/alcohol screen.
* Positive human immunodeficiency virus (HIV) antibody test.
* Positive coronavirus disease 2019 (COVID-19): SARS-CoV2 polymerase chain reaction (PCR) or lateral flow test of a combined throat and nasopharyngeal swab or nasal swab only.
* Regular alcohol consumption within 6 months prior to the study defined as: an average weekly intake of >14 units for males and >14 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Regular use of known drugs of abuse.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates participation in the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Australia (2):
  - GSK Investigational Site, Herston Queensland, Queensland
  - GSK Investigational Site, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 91 participants screened, 32 participants were enrolled in the study (57 participants were screen failures). The most common reasons for screen failure were not meeting inclusion/exclusion criteria for 45 participants and physician decision for 10 participants.
Pre-assignment Details: Of 32 participants who were enrolled and randomized, 1 participant from GSK3858279 Caucasian arm did not receive any study intervention due to high blood pressure (BP). A total of 29 participants completed the study (Placebo: 10 participants [91%] and GSK3858279: 19 participants [95%]).
Period: Overall Study
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Started | 6 | 7 | 7 | 4 | 3 | 4
Completed | 6 | 7 | 6 | 3 | 3 | 4
Not Completed | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSK3858279 Caucasian: Participants received 240 mg of GSK3858279 administered as separate subcutaneous (SC) injection to healthy Caucasian participants.
- Total: Total of all reporting groups
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo | Total
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4 | 31
Age, Customized [Count of Participants; unit: Participants] — The Age of the participants was measured in Years of life.
  Participants
    20 - 65 (years of age) | 6 | 7 | 7 | 4 | 3 | 4 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Male | 6 | 7 | 7 | 3 | 3 | 4 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN | 0 | 7 | 7 | 0 | 3 | 4 | 21
  WHITE | 6 | 0 | 0 | 4 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants With Adverse Events (AEs), Serious Adverse Events (SAE's) And Withdrawals Due to AE's
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAEs are defined as any untoward medical occurrence that, at any dose: results in death, cause life threatening events which requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability or incapacity and birth defect or congenital anomaly. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169.
Time Frame: Up to 169 days
Population: The analysis was performed on the Safety Set that included all randomized participants who received at least one injection of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Participants
  AE | 5 | 6 | 2 | 4 | 1 | 2
  SAE | 0 | 0 | 0 | 0 | 0 | 0
  Withdrawals Due to AE | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Hematology Parameter of Platelet Count
Description: Blood samples were collected for the assessment of change from baseline in hematology parameter platelet count. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Giga cells per liter (10^9/L) | 2.8 (25.90) | 18.0 (18.81) | -4.2 (12.27) | 7.0 (15.59) | 16.0 (39.60) | -12.3 (6.51)

3. Primary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters Hemoglobin. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gram Per Liter (g/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Gram Per Liter (g/L) | -7.5 (13.79) | -6.0 (10.42) | -2.0 (10.79) | -5.3 (7.37) | -10.5 (16.26) | -3.0 (3.61)

4. Primary Outcome: Change From Baseline in Hematology Parameter of Hematocrit
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters Hematocrit. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter/liter (L/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Liter/liter (L/L) | -0.027 (0.0367) | -0.010 (0.0408) | -0.005 (0.0259) | -0.027 (0.0321) | -0.035 (0.0495) | -0.013 (0.0208)

5. Primary Outcome: Change From Baseline in White Blood Cell (Wbc) Count With Differential i.e. Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Blood samples were collected for the assessment of hematology parameters including (WBC) count with differential i.e. Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: The analysis was performed on the Safety Set that included all randomized participants who received at least one injection of study intervention. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 2 | 5 | 3 | 2 | 3
Giga cells per liter (10^9/L)
  Basophils: number analyzed (Participants) | 6 | 2 | 4 | 1 | 2 | 3
  Basophils | 0.01 (0.020) | 0.00 (0.000) | 0.00 (0.000) | 0.00 (0.00) | -0.03 (0.035) | 0.00 (0.000)
  Eosinophils | 0.00 (0.084) | -0.03 (0.035) | 0.02 (0.135) | -0.07 (0.115) | 0.03 (0.035) | 0.68 (1.098)
  Lymphocytes | 0.02 (0.172) | 0.10 (0.141) | 0.04 (0.261) | 0.03 (0.306) | 0.15 (0.212) | -0.20 (0.361)
  Monocytes | 0.00 (0.063) | 0.05 (0.071) | 0.10 (0.122) | -0.10 (0.265) | 0.05 (0.071) | 0.10 (0.100)
  Neutrophils | -0.12 (0.791) | -0.25 (0.212) | 0.54 (1.001) | -0.97 (1.079) | 1.15 (1.061) | 0.07 (0.462)

6. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP)
Description: Blood samples were collected for the assessment of clinical chemistry parameters including AST, ALT, AP. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 2 | 3
Units per liter (U/L)
  Alkaline Phosphatase (AP) | 0.8 (12.16) | 1.3 (6.34) | -6.5 (14.18) | 0.0 (7.94) | -3.0 (8.49) | -4.3 (11.06)
  Alanine Aminotransferase (ALT) | 3.2 (9.70) | 9.3 (17.25) | 4.0 (4.15) | 17.3 (5.13) | -3.0 (5.66) | -2.0 (11.79)
  Aspartate Aminotransferase (AST) | 2.3 (5.72) | 12.0 (19.37) | 0.8 (6.74) | 11.0 (3.61) | 1.0 (4.24) | -1.3 (3.06)

7. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Protein
Description: Blood samples were collected for the assessment of clinical chemistry parameters including total Protein. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Gram Per Liter (g/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Gram Per Liter (g/L) | 2.2 (1.94) | 2.5 (2.89) | 0.8 (4.45) | 0.3 (2.52) | -0.5 (4.95) | 3.3 (1.53)

8. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin
Description: Blood samples were collected for the assessment of clinical chemistry parameters including Total bilirubin. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: micromole per liter (umol/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
micromole per liter (umol/L) | -5.3 (3.88) | -0.3 (4.79) | -1.5 (3.73) | -4.7 (1.53) | 0.5 (2.12) | 1.3 (6.03)

9. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Direct Bilirubin, Creatinine
Description: Blood samples were collected for the assessment of clinical chemistry parameters including Direct bilirubin, Creatinine. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: micromole per liter (umol/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 2 | 3
micromole per liter (umol/L)
  Direct Bilirubin, | -1.8 (1.47) | 0.0 (2.16) | -0.3 (0.82) | -1.7 (0.58) | 0.0 (1.41) | 1.3 (3.51)
  Creatinine | 1.8 (8.86) | -1.8 (8.85) | 3.0 (4.94) | 5.7 (10.69) | 14.5 (7.78) | 0.0 (3.61)

10. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter of Urea, Glucose, Potassium, Sodium
Description: Blood samples were collected for the assessment of clinical chemistry parameters including Urea, Glucose, Potassium, Sodium. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 2 | 3
millimoles per liter (mmol/L)
  Glucose | 0.25 (0.575) | 0.03 (0.171) | 0.18 (0.549) | 0.23 (0.651) | 1.10 (1.980) | 0.27 (0.208)
  Potassium | 0.00 (0.400) | -0.08 (0.189) | -0.15 (0.302) | 0.33 (0.115) | -0.45 (0.212) | 0.03 (0.058)
  Sodium | 1.8 (0.98) | -1.8 (3.40) | 0.5 (3.02) | 0.7 (1.53) | 0.0 (1.41) | 1.0 (0.00)
  Urea | 1.43 (0.907) | 0.38 (1.715) | 0.87 (1.718) | 1.03 (0.862) | 1.45 (0.495) | 1.13 (0.723)

11. Primary Outcome: Number of Participants With Change From Baseline in Urinalysis Parameter: Urine Specific Gravity (Ratio of Urine Density to Water Density)
Description: Urine samples were collected to analyze the urinalysis parameter: specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine, indicated as ratio of urine density to water density. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Participants
  Any Increase | 6 | 7 | 7 | 4 | 3 | 4
  Increase to 1.019 | 0 | 0 | 1 | 0 | 0 | 0
  Increase to 1.02 | 1 | 0 | 0 | 0 | 0 | 0
  Increase to 1.021 | 1 | 0 | 0 | 1 | 0 | 0
  Increase to 1.024 | 0 | 0 | 2 | 0 | 0 | 0
  Increase to 1.025 | 1 | 1 | 0 | 1 | 0 | 0
  Increase to 1.026 | 0 | 0 | 0 | 1 | 0 | 0
  Increase to 1.027 | 0 | 0 | 0 | 0 | 1 | 0
  Increase to 1.028 | 0 | 1 | 0 | 1 | 0 | 0
  Increase to 1.029 | 1 | 0 | 0 | 0 | 0 | 1
  Increase to 1.03 | 0 | 3 | 0 | 0 | 1 | 0
  Increase to 1.031 | 0 | 0 | 1 | 0 | 0 | 0
  Increase to 1.032 | 0 | 0 | 1 | 0 | 1 | 2
  Increase to 1.033 | 0 | 1 | 1 | 0 | 0 | 1
  Increase to 1.034 | 1 | 0 | 1 | 0 | 0 | 0
  Increase to 1.036 | 1 | 1 | 0 | 0 | 0 | 0

12. Primary Outcome: Number of Participants With Change From Baseline in Urinalysis Parameter: Urine Potential of Hydrogen (pH)
Description: Urine samples were collected to analyze the urinalysis parameter: pH. Urine pH is an acid-base measurement. pH is measured on a numeric scale ranging from 0 to 14; values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH less than 7 is acidic, and a pH greater than 7 is basic. Normal urine has a slightly acidic pH (5.0 - 6.0). The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated as post-dose visit value minus the Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Participants
  Any Increase | 5 | 6 | 4 | 2 | 2 | 3
  Increase to 6.5 | 1 | 2 | 0 | 0 | 0 | 0
  Increase to 7.0 | 1 | 0 | 0 | 0 | 0 | 1
  Increase to 7.5 | 1 | 2 | 2 | 0 | 2 | 2
  Increase to 8.0 | 1 | 2 | 2 | 2 | 0 | 0
  Increase to 8.5 | 1 | 0 | 0 | 0 | 0 | 0

13. Primary Outcome: Number of Participants With Abnormal Urinalysis Results by Dipstick Method
Description: The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameters can be read as increase to trace, increase to 1+ (low concentrations present), increase to 2+ (moderate concentrations present) and increase to 3+ (high concentrations present) indicating proportional concentrations in the urine sample. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Data for worst-case post-Baseline relative to Baseline is presented.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Participants
  Bilirubin, Any Increase | 1 | 1 | 1 | 0 | 0 | 0
  Bilirubin, Increase to TRACE | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Increase to 1+ | 1 | 1 | 1 | 0 | 0 | 0
  Bilirubin, Increase to 2+ | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Increase to 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Bilirubin, Increase to 4+ | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Any Increase | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Increase to TRACE | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Increase to 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Increase to 2+ | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Increase to 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, Increase to 4+ | 0 | 0 | 0 | 0 | 0 | 0
  Ketones, Any Increase | 3 | 5 | 4 | 2 | 3 | 1
  Ketones, Increase to TRACE | 3 | 5 | 3 | 2 | 3 | 1
  Ketones, Increase to 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Ketones, Increase to 2+ | 0 | 0 | 1 | 0 | 0 | 0
  Ketones, Increase to 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Ketones, Increase to 4+ | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte Esterase, Any Increase | 0 | 0 | 0 | 1 | 0 | 1
  Leukocyte Esterase, Increase to TRACE | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte Esterase, Increase to 1+ | 0 | 0 | 0 | 1 | 0 | 1
  Leukocyte Esterase, Increase to 2+ | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte Esterase, Increase to 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Leukocyte Esterase, Increase to 4+ | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite, Any Increase | 0 | 0 | 0 | 0 | 0 | 0
  Nitrite, Increase to POSITIVE | 0 | 0 | 0 | 0 | 0 | 0
  Occult Blood, Any Increase | 1 | 1 | 1 | 1 | 0 | 0
  Occult Blood, Increase to TRACE | 0 | 1 | 0 | 0 | 0 | 0
  Occult Blood, Increase to 1+ | 1 | 0 | 1 | 0 | 0 | 0
  Occult Blood, Increase to 2+ | 0 | 0 | 0 | 1 | 0 | 0
  Occult Blood, Increase to 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Occult Blood, Increase to 4+ | 0 | 0 | 0 | 0 | 0 | 0
  Protein, Any Increase | 2 | 2 | 2 | 1 | 0 | 2
  Protein, Increase to TRACE | 2 | 1 | 2 | 1 | 0 | 2
  Protein, Increase to 1+ | 0 | 1 | 0 | 0 | 0 | 0
  Protein, Increase to 2+ | 0 | 0 | 0 | 0 | 0 | 0
  Protein, Increase to 3+ | 0 | 0 | 0 | 0 | 0 | 0
  Protein, Increase to 4+ | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen, Any Increase | 0 | 0 | 1 | 0 | 0 | 0
  Urobilinogen, Increase to TRACE | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen, Increase to 1+ | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen, Increase to 2+ | 0 | 0 | 0 | 0 | 0 | 0
  Urobilinogen, Increase to 3+ | 0 | 0 | 1 | 0 | 0 | 0
  Urobilinogen, Increase to 4+ | 0 | 0 | 0 | 0 | 0 | 0

14. Primary Outcome: Change From Baseline in Vital Signs: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: The vital sign followed in this analysis was both systolic and diastolic blood pressure, expressed as millimetre of mercury. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Millimetre of Mercury (mmHg)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 2 | 3
Millimetre of Mercury (mmHg)
  Systolic Blood Pressure | 5.3 (13.00) | 0.8 (7.37) | 0.8 (6.18) | -1.0 (7.21) | 5.0 (5.66) | 0.0 (5.00)
  Diastolic Blood Pressure | 5.2 (10.26) | 4.0 (2.00) | 3.5 (8.24) | 1.3 (4.73) | 8.5 (12.02) | -1.0 (3.61)

15. Primary Outcome: Change From Baseline in Vital Signs: Pulse Rate
Description: The vital signs followed in this analysis was pulse rate, expressed as beats per minute. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Beats per minute (bpm) | 6.5 (11.74) | 16.0 (18.17) | 6.8 (11.58) | 6.7 (6.03) | 10.0 (1.41) | 4.3 (9.02)

16. Primary Outcome: Change From Baseline in Vital Signs: Body Temperature
Description: The vital sign followed in this analysis was body temperature, expressed as degree Celsius. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Degree Celsius | 0.07 (0.468) | -0.03 (0.330) | 0.48 (0.436) | -0.10 (0.500) | 0.00 (0.141) | -0.03 (0.115)

17. Primary Outcome: Change From Baseline in Vital Signs: Respiratory Rate
Description: The vital signs followed in this analysis was respiratory rate, expressed as Breaths per minute. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Change from Baseline was defined as value at the indicated time point minus Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Breaths per minute | -0.5 (1.76) | -0.8 (0.96) | -1.0 (1.67) | -2.0 (2.00) | -0.5 (2.12) | -0.7 (2.31)

18. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters: PR Interval, QRS Duration, QT Interval and QT Interval Corrected for Heart Rate According to Fridericia's Formula (QTcF) Interval
Description: Twelve-lead ECG were obtained to measure PR Interval, QRS Duration, QT Interval, QTcF Interval and QTcB Interval. Twelve-lead ECGs were performed with the participant in a supine or semi-supine position after a rest of at least 10 minutes. The final follow-up visit was on Day 169 for participants in the Caucasian cohort and on Day 113 for Chinese and Japanese participants respectively (NB: Japanese and Chinese participants had an option to remain in the study until Day 169). Baseline was defined as the average of the triplicate pre-dose assessments on Day 1 of Period 2. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline and Day 169
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 4 | 6 | 3 | 2 | 3
milliseconds (msec)
  PR Interval | -5.000 (6.4601) | -4.000 (7.4486) | -7.889 (21.1152) | -15.778 (7.5817) | -8.167 (4.4783) | 6.111 (12.6242)
  QRS Duration | -2.833 (7.9631) | -2.083 (4.7561) | -0.444 (8.8410) | 1.667 (6.2272) | 3.167 (3.5355) | -3.667 (4.5092)
  QT Interval | -16.278 (26.0431) | -7.083 (15.8052) | -18.056 (33.7859) | -15.222 (16.4057) | -21.333 (26.8701) | -7.111 (14.6148)
  QTcB Interval | 4.333 (12.5131) | 5.917 (8.7575) | 7.333 (8.8292) | 13.667 (9.5975) | 21.500 (17.2063) | -2.444 (7.1518)
  QTcF Interval | -2.333 (13.5859) | 1.583 (4.9319) | -2.611 (15.3122) | 3.778 (11.4956) | 6.667 (20.2704) | -4.111 (9.7144)

19. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 56 Days AUC (0-56)] of GSK3858279
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate pharmacokinetic (PK) parameters. PK parameter population consist of all participants in the PK Population, for whom valid and evaluable PK parameters were derived. This population was used in the assessment and characterization of PK parameters.
Time Frame: Predose, 6 Hour (h), 12 h, 24 h, 36 h, 48 h (post dose till Day 3), Day 8, 15, 22, 29, 43 and 57
Population: All participants in the safety population who received an active dose of study treatment and had at least one reportable Pharmacokinetic (PK) assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day* nanograms per milliliter (ng/mL)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese
Number analyzed (Participants) | 6 | 7 | 7
day* nanograms per milliliter (ng/mL) | 87592.7 (15.8) | 86412.2 (28.2) | 77742.0 (22.5)

20. Primary Outcome: AUC From Time Zero to the Last Measurable Concentration (0-t) Post-Dose of GSK3858279
Description: as for outcome 19
Time Frame: Predose, 6 Hour (h), 12 h, 24 h, 36 h, 48 h (post dose till Day 3), Day 8, 15, 22, 29, 43, 57, 85, 113, 141, 155 and 169 Days
Population: All participants in the safety population who received an active dose of study treatment and had at least one reportable PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*nanograms per milliliter (day*ng/mL)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese
Number analyzed (Participants) | 6 | 7 | 7
day*nanograms per milliliter (day*ng/mL) | 88679.6 (17.6) | 87201.8 (29.1) | 77009.4 (21.0)

21. Primary Outcome: Time of Occurrence of Last Quantifiable Concentration (Tlast) of GSK3858279
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Median (Full Range); unit: day
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese
Number analyzed (Participants) | 6 | 7 | 7
day | 56.115 [41.83 to 84.92] | 56.062 [54.93 to 84.06] | 55.964 [14.01 to 58.01]

22. Primary Outcome: Maximum Observed Concentration (Cmax) of GSK3858279
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese
Number analyzed (Participants) | 6 | 7 | 7
nanograms per milliliter (ng/mL) | 9135.3 (42.0) | 6851.4 (41.4) | 8295.4 (39.8)

23. Primary Outcome: Time of Occurrence of Cmax (Tmax) of GSK3858279
Description: as for outcome 21
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Median (Full Range); unit: day
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese
Number analyzed (Participants) | 6 | 7 | 7
day | 2.004 [1.50 to 7.03] | 3.919 [1.50 to 7.18] | 3.217 [1.00 to 4.15]

24. Secondary Outcome: Percentage Change From Baseline in Free CCL17
Description: Blood samples were collected from participants at time points after the administration of study treatment to investigate PK parameters. The study intervention dose was administered on Study Day 1(baseline), where 7 days post-dose totals to Study Day 1+7days = Study Day 8. Following results of Day 8, Day 15, Day 29 and Day 57 corelates to timepoints Day 7, Day 14, Day 28 and Day 56 post dose values and same are presented here.
Time Frame: Baseline (Day 1) and at Days 7, 14, 28 and 56 Post dose
Population: All participants in the safety population who had at least one reportable Target Engagement (TE) assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change (%)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Percent change (%)
  Day 8, Percent change | 89.715 [87.619 to 91.490] | 85.825 [81.308 to 89.393] | 88.461 [83.293 to 92.181] | 22.353 [7.695 to 49.851] | 0.452 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.863 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values.
  Day 15, Percent change: number analyzed (Participants) | 5 | 7 | 7 | 4 | 3 | 4
  Day 15, Percent change | 60.524 [46.235 to 73.216] | 50.249 [34.215 to 66.232] | 59.183 [44.561 to 72.343] | 7.528 [0.067 to 90.873] | 0.528 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.787 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values.
  Day 29, Percent change: number analyzed (Participants) | 6 | 7 | 6 | 3 | 3 | 4
  Day 29, Percent change | 0.529 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.165 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.606 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 3.665 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.316 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.558 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values.
  Day 57, Percent change: number analyzed (Participants) | 6 | 7 | 6 | 4 | 3 | 4
  Day 57, Percent change | 1.380 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.100 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 0.527 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 14.136 [1.811 to 59.507] | 1.416 [NA to NA] — Free CCL17 values below the Lower limit of quantification (LLQ) are imputed to be (1/2) *LLQ = 0.1. If more than 30% of values have been imputed at any timepoint for a treatment group, then CI has not been calculated due to the high proportion of non-quantifiable (NQ) values that have been imputed which may affect the CI values. | 2.875 [0.069 to 55.775]

25. Secondary Outcome: Cmax of Total CCL17 in Serum Following GSK3858279
Description: as for outcome 21
Time Frame: Baseline (Day 1) and at Days 7, 14, 28 and 56 Post dose
Population: All participants in the safety population who had at least one reportable TE assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter (pg/mL)
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Picogram per milliliter (pg/mL) | 68969.794 (30.025) | 62648.760 (29.529) | 55177.740 (20.370) | 1661.847 (31.284) | 733.904 (4.084) | 621.421 (61.396)

26. Secondary Outcome: Tmax of Total CCL17 in Serum Following GSK3858279
Description: Blood samples were collected from participants at indicated time points after the administration of study treatment to investigate PK parameters. The study intervention dose was administered on Study Day 1(baseline), where 7 days post-dose totals to Study Day 1+7days = Study Day 8. Following results of Day 8, Day 15, Day 29 and Day 57 corelates to timepoints Day 7, Day 14, Day 28 and Day 56 post dose values and same are presented here.
Time Frame: Baseline (Day 1) and at Days 7, 14, 28 and 56 Post dose
Population: All participants in the safety population who had at least one reportable TE assessment.
Measure: Mean (Standard Deviation); unit: day
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
day | 9.333 (5.7155) | 14.000 (4.0415) | 8.571 (3.8668) | 57.000 (75.7276) | 1.083 (0.7217) | 26.313 (38.8659)

27. Secondary Outcome: Maximum Fold Change in Total CCL17 in Serum Following GSK3858279 Administration
Description: as for outcome 21
Time Frame: Baseline (Day 1) and Days 56 Post dose
Population: All participants in the safety population who had at least one reportable TE assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Fold Change
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Fold Change | 77.479 (4.674) | 113.436 (34.212) | 73.474 (58.664) | 1.155 (14.377) | 1.270 (3.027) | 1.383 (29.136)

28. Secondary Outcome: Fold Increase in Total CCL17 in Serum Following GSK3858279 Administration
Description: as for outcome 26
Time Frame: Baseline (Day 1) and at Days 7, 14, 28 and 56 Post dose
Population: All participants in the safety population who had at least one reportable TE assessment.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Change
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Fold Change
  Day 8 | 76.489 [70.870 to 82.552] | 93.537 [76.813 to 113.903] | 70.025 [42.278 to 115.981] | 0.866 [0.689 to 1.089] | 0.975 [0.750 to 1.268] | 1.025 [0.730 to 1.439]
  Day 15 | 61.874 [51.206 to 74.765] | 110.634 [81.785 to 149.659] | 56.857 [27.424 to 117.878] | 0.977 [0.678 to 1.409] | 1.000 [0.798 to 1.254] | 1.072 [0.819 to 1.403]
  Day 29 | 26.405 [22.124 to 31.515] | 61.250 [46.002 to 81.552] | 21.448 [9.707 to 47.388] | 0.971 [0.495 to 1.904] | 0.960 [0.881 to 1.046] | 1.145 [0.858 to 1.528]
  Day 57 | 7.049 [4.323 to 11.495] | 16.002 [11.436 to 22.391] | 5.056 [2.583 to 9.894] | 0.942 [0.682 to 1.301] | 0.867 [0.745 to 1.009] | 1.082 [0.798 to 1.468]

29. Secondary Outcome: Number of Participants With Pre-existing Anti-drug Antibodies (ADA's)
Description: Serum samples were collected for the determination of anti- GSK3858279 antibodies (ADA). The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample. Additionally, confirmed positive ADA samples were also tested in a validated neutralizing antibody assay to determine the potential neutralizing activity of the ADA.
Time Frame: Day 169
Population: All participants in the safety population who had at least one reportable TE assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

30. Secondary Outcome: Number of Participants With Treatment-Emergent ADA's Over Time
Description: Serum samples were collected for the determination of anti- GSK3858279 antibodies (ADA).The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample. Additionally, confirmed positive ADA samples were also tested in a validated neutralizing antibody assay to determine the potential neutralizing activity of the ADA.
Time Frame: Day 169
Population: All participants in the safety population who had at least one reportable TE assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
Number analyzed (Participants) | 6 | 7 | 7 | 4 | 3 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected from the start of the study intervention up to Day 169.
Description: All-cause mortality, Serious adverse events and non-serious adverse events were reported for the Safety Population who were randomized and received at least one dose of study
Arm/Group | GSK3858279 Caucasian | GSK3858279 Chinese | GSK3858279 Japanese | Caucasian Placebo | Chinese Placebo | Japanese Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7 | 0/7 | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/7 | 0/4 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 5/6 | 6/7 | 2/7 | 4/4 | 1/3 | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3858279 Caucasian (N=6) | GSK3858279 Chinese (N=7) | GSK3858279 Japanese (N=7) | Caucasian Placebo (N=4) | Chinese Placebo (N=3) | Japanese Placebo (N=4)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/13/NCT05174013/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/13/NCT05174013/SAP_001.pdf